CLINICAL TRIAL: NCT01100541
Title: Evaluation of a Polymeric Plate Derived From Castor Oil to Thermotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Fabiula Barbosa Machado dos Santos, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CEPHCFMRPUSP-11099
Record Dates: First submitted 2010-04-06; First posted 2010-04-09 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Therapeutic Hyperthermia; Thermotherapy; Polymers
Keywords: Therapeutic Hyperthermia; Thermotherapy; Polymers; Castor Oil
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Polymeric plate characteristics (Experimental): Evaluation, in the volunteers viewpoint, of the polymeric plate characteristics.
  Interventions: Device: Polymeric plate

INTERVENTIONS:
Device: Polymeric plate — Application of the polymeric plate in the shoulder for 20 minutes after warming it for 15 minutes in hot water, initially at boiling temperature.
  Other Names: PPDOM; PPDCO

SUMMARY:
The objective of this work is to evaluate, from volunteers viewpoint, the usability, comfort, appearance, weight, superficial temperature, and other characteristics of a polymeric plate derived from castor oil developed to thermotherapy.

The volunteers will use polymeric plate as a therapeutic resource in the shoulder area and then fill in, without interference of the researcher, some questions about the characteristics of interest.

DETAILED DESCRIPTION:
In this study, the polymeric plate is prepared using the following procedure:

1. - the water is heated to the boiling temperature
2. - the heater is shut down
3. - the polymeric plate is immersed in water
4. - it rests in the water for 15 minutes
5. - it is inserted in a wrap

In this condition, the polymeric plate is placed on the shoulder of the volunteer and remains there for 20 minutes.

After application, the volunteer answers the questionnaire containing eight questions on a Likert scale (0 to 10) and an area of observations.

Previous laboratory tests were performed to ensure that the temperature of the polymeric plate will not cause skin burn in this application condition.

ELIGIBILITY:
Inclusion Criteria:

* Good communication and comprehension
* Skin integrity

Exclusion Criteria:

* Reduced skin sensitivity
* Disturbance in the central nervous system

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Acceptance of the polymeric plate | 2 weeks
  Acceptance of the polymeric plate by the volunteers.

SECONDARY OUTCOMES:
Polymeric plate comfort | 2 weeks
  Perception of the volunteers about the comfort of the polimeric plate.
Polymeric plate temperature | 2 weeks
  Perception of the volunteers about the polymeric plate temperature.
Polymeric plate time of heat retention | 2 weeks
  Perception of the volunteers about the polymeric plate time of heat retention.
Sensation on the superficial touch of the polymeric plate | 2 weeks
  Perception of the volunteers about the sensation on the superficial touch of the polymeric plate.
Appearance of the polymeric plate | 2 weeks
  Perception of the volunteers about the appearence of the polymeric plate.
Polymeric plate weight | 2 weeks
  Perception of the volunteers about the polymeric plate weight.
Polymeric plate practicality | 2 weeks
  Perception of the volunteers about the polymeric plate practicality.
General observations about the polymeric plate | 2 weeks
  General comments, suggestions and complaints of the volunteers about the polymeric plate.

CONTACTS AND LOCATIONS:
Overall Officials: Fabiula BM dos Santos, Physio, Principal Investigator — University of Sao Paulo; Valéria MC Elui, PhD, Study Director — University of Sao Paulo
Locations (1):
- Interunits postgraduate program in bioengineering, São Carlos, São Paulo, Brazil